CLINICAL TRIAL: NCT02081677
Title: One Month Daily Wear Clinical Evaluation of Three Prototype Soft Contact Lenses in a Population of Habitual and Neophyte Contact Lens Wearers
Brief Title: One Month Daily Wear Clinical Evaluation of New Prototype Contact Lenses in Habitual and Neophyte Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5146
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-07

CONDITIONS: Visual Correction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- etafilcon A (Active Comparator): Marketed control soft contact lens
  Interventions: Device: ACUVUE 2
- Prototype E1 (Experimental): Investigational soft contact lens
  Interventions: Device: Prototype E1
- Prototype E2 (Experimental): Investigational soft contact lens
  Interventions: Device: Prototype E2
- Prototype E3 (Experimental): Investigational soft contact lens
  Interventions: Device: Prototype E3

INTERVENTIONS:
Device: ACUVUE 2 — worn in a daily wear modality; lenses will be replaced after 2 weeks
  Arms: etafilcon A
Device: Prototype E1 — worn in a daily wear modality; lenses will be replaced after 2 weeks
  Other Names: Investigational soft contact lens
  Arms: Prototype E1
Device: Prototype E2 — worn in a daily wear modality; lenses will be replaced after 2 weeks
  Other Names: Investigational soft contact lens
  Arms: Prototype E2
Device: Prototype E3 — worn in a daily wear modality; lenses will be replaced after 2 weeks
  Other Names: Investigational soft contact lens
  Arms: Prototype E3

SUMMARY:
There will be four study lenses tested; one marketed lens, and three prototype study lenses. Subjects will be randomized to one of the four study lenses which will be worn in a daily wear modality, with a two week replacement.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be between 18 and 39 years of age.
2. The subject must be able to read and understand English.
3. The subject read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form.
4. The subject must not have been a participant in a contact lens or contact lens solution study/investigation in the previous seven days.
5. The subject must be willing to wearthe study lenses for at least 6 hours per day, 7 days per week (e.g. does not regularly swim).
6. The subject must appear able and willing and able to the adhere to the instructions set forth in this clinical protocol.
7. The subject's subjective refraction must result in a vertex corrected spherical contact lens prescription in the range of -1.00D to -4.00D in each eye.
8. The subject's refractive astigamatism must be less than or equal to -1.00D in both eyes.
9. The subjet must have best corrected visual acuity of 20/30 (6/9 or +0.20 logMAR) or better in each eye.
10. The subject must require a visual correction in both eyes (no monofit or monovision allowed).
11. The subject must have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

    * No amblyopia
    * No evidence of lid abnormality or infection (including blepharitis/meibomitis)
    * No conjunctival abnormality or infection.
    * No clinically significant slit lamp findings (i.e. stromal edema, vascularization, corneal scaring, infiltrates or abnormal opacities).
    * No other active ocular diseases.

Exclusion Criteria:

1. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
2. Any systemic diseases, autoimmune disease, or use of medication, which may interfere with contact lens wear.
3. Clinically significant (Grade 3 or 4) corneal edeam, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
4. Any ocular infection.
5. Any corneal distortion resulting from previous hard or rigid permeable contact lens wear.
6. Pregnancy or lactation (subjects who become pregnant during the study will be discontinued).
7. No extended wear in the last 3 months.
8. Diabetes.
9. Infectious diseases (e.g. hepatitis, tuberculosis) or immunosuppressive disease (e.g. HIV).
10. Has had refractive surgery.
11. Employee of VRF with direct involvement in the study or a family member of the clinic.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2014-06-25 (Actual); Study Completion 2014-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chennai, Tamil Nadu, India

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 80 subjects were enrolled in this study. Of the enrolled subjects 4 did not meet the eligibility criteria and 76 were randomized to receive a study lens. Of the randomized subjects 72 completed the study.
Groups:
- Etafilcon A: Subjects that were randomized to receive etafilcon A contact lens throughout the course of this study.
- Prototype E1: Subjects that were randomized to receive Prototype E1 contact lens throughout the course of this study.
- Prototype E2: Subjects that were randomized to receive Prototype E2 contact lens throughout the course of this study.
- Prototype E3: Subjects that were randomized to receive Prototype E3 contact lens throughout the course of this study.
Period: Overall Study
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Started | 19 | 19 | 19 | 19
Completed | 18 | 18 | 17 | 19
Not Completed | 1 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 1 | 0
Not completed — Not comfortable with lens care system | 1 | 0 | 0 | 0
Not completed — Unsatisfactory Lens Fitting | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were enrolled into the study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3 | Total
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.42 (4.611) | 24.58 (4.706) | 23.16 (5.336) | 20.84 (2.192) | 23.0 (4.211)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 11 | 11 | 48
  Male | 7 | 5 | 8 | 8 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Asian Indian | 19 | 19 | 19 | 19 | 76
Region of Enrollment [Number; unit: participants]
  India | 19 | 19 | 19 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining (Area)
Description: Corneal Staining Area was collected at baseline and 4- week evaluations in both eyes using a slit lamp and was graded with a 11-point scale (i.e. Grade 0= 0% of region covered, Grade 1 =10% of region covered, Grade 2 = 20% of region covered, Grade 3 = 30% of region covered, Grade 4= 40% of region covered, Grade 5 = 50% of region covered, Grade 6 = 60% of region covered,Grade 7 = 70% of region covered, Grade 8 = 80% of region covered, Grade 9 = 90% of region covered and Grade 10 = 100% of region covered). Central, interior, nasal, temporal and superior locations were evaluated. The average grade for each lens and time point was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: The analysis population consist of all subjects that completed all study visits without a major protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Units on a scale
  Baseline | 11.76 (24.676) | 5.79 (18.4) | 4.17 (6.918) | 6.18 (17.925)
  4-week Follow-up | 5.29 (12.367) | 4.21 (9.482) | 8.06 (7.491) | 9.69 (8.224)

2. Primary Outcome: Corneal Staining (Depth)
Description: Corneal Staining Depth was collected at baseline and 4- week evaluations in both eyes using a slit lamp and was graded with a 4-point scale (i.e. Grade 0= None, Grade 1 =Superficial epithelial, Grade 2 = Full epithelial, Grade 3 =stromal glow). Central, interior, nasal, temporal and superior locations were evaluated. The average grade for each lens and time point was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: The analysis population consist of all subjects that completed all study visits without a major protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Units on a scale
  Baseline | 1.03 (2.037) | 0.45 (1.224) | 0.36 (0.593) | 0.44 (1.045)
  4-week Follow-up | 0.53 (1.237) | 0.42 (0.948) | 0.81 (0.749) | 0.97 (0.822)

3. Primary Outcome: Corneal Staining (Type)
Description: Corneal Staining was collected at baseline and 4- week evaluations in both eyes using a slit lamp and was graded with a 5-point scale (i.e. Grade 0= None, Grade 1 =Micropunctate, Grade 2 = Macropunctate, Grade 3 = Coalesced Macropunctate and Grade 4 = Patch (greater or equal to 1mm). Central, interior, nasal, temporal and superior locations were evaluated. The average grade for each lens and time point was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: The analysis population consist of all subjects that completed all study visits without a major protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Units on a scale
  Baseline | 1.03 (2.037) | 0.58 (1.840) | 0.42 (0.692) | 0.59 (1.829)
  4-week Follow-up | 0.53 (1.237) | 0.42 (0.948) | 0.81 (0.749) | 0.94 (0.801)

4. Primary Outcome: Limbal Conjunctival Redness
Description: Limbal Conjunctival Redness was assessed for each subject and eye at baseline and 2-week follow-up evaluations. Limbal Redness was assessed in 4 regions Inferior, Nasal, Temporal and Superior and Graded using an Efron Grading scale for limbal redness in 0.5 unit increments (Grade 0:None, Grade 1:Trace, Grade 2: Mild, Grade 3: Moderate and Grade 4: Severe). The average Grade across all four regions can range from 0 to 16 where lower values indicate better performance. The average Grade for each individual region can range from 0 to 4. The average grade across all regions was reported for each lens and time point.
Time Frame: Baseline and 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Subject Eye
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eye) | 34 | 38 | 36 | 32
units on a scale
  Baseline | 4.0 (1.822) | 3.50 (1.564) | 3.72 (1.485) | 4.06 (1.294)
  2-week Follow-up | 3.93 (1.441) | 3.54 (1.472) | 3.72 (1.446) | 3.53 (1.646)

5. Primary Outcome: Bulbar Conjunctival Redness
Description: Bulbar Conjunctival Redness was assessed for each subject and eye at baseline and 2-week follow-up evaluations. Bulbar Redness was assessed in 4 regions Inferior, Nasal, Temporal and Superior and Graded using an Efron Grading scale for bulbar redness in 0.5 unit increments (Grade 0:None, Grade 1:Trace, Grade 2: Mild, Grade 3: Moderate and Grade 4: Severe). The average Grade across all four regions can range from 0 to 16 where lower values indicate better performance. The average Grade for each individual region can range from 0 to 4. The average grade across all regions was reported for each lens and time point.
Time Frame: Baseline and 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Subject Eye
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eye) | 34 | 38 | 36 | 32
units on a scale
  Baseline | 4.04 (1.378) | 4.12 (1.416) | 4.08 (1.099) | 4.24 (1.136)
  2-week Follow-up | 4.13 (1.170) | 4.47 (0.870) | 4.18 (1.166) | 4.28 (1.431)

6. Primary Outcome: Visual Acuity (LogMAR)
Description: Visual Acuity (LogMAR) was assessed bionocularly at the 4-week follow-up evaluations. The average visual acuity (LogMAR) for each lens was reported.
Time Frame: 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
LogMAR | -0.15 (0.078) | -0.12 (0.067) | -0.13 (0.076) | -0.13 (0.086)

7. Primary Outcome: Lens Fitting Characteristics
Description: Lens fit was assessed for each subject eye at post lens fitting and 4- week follow-up evaluations. Lens fit is a binary response as acceptable or unacceptable lens fit. The percentage of eyes with acceptable lens fit was reported.
Time Frame: Post Lens Fitting and 4-Week Follow-up
Population: The analysis population consists of all subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Post Lens Fitting | 100 | 100 | 100 | 100
  4-week Follow-up | 100 | 100 | 100 | 100

8. Primary Outcome: Percentage of Reported Ocular Symptoms (Burning/Stinging)
Description: The Ocular symptom Burning/Stinging was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 5.9 | 0.0 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 6.3

9. Primary Outcome: Corneal Edema
Description: Corneal Edema was assessed using a bio-microscope at baseline and 4- week evaluations in both eyes and was graded with a 5-point scale (Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). The Percentage of eyes with Grade 3 or higher was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0 | 0 | 0 | 0
  4-week Follow-up | 0 | 0 | 0 | 0

10. Primary Outcome: Conjunctival Injection
Description: Conjunctival Injection was assessed using a bio-microscope at baseline and 4- week evaluations in both eyes and was graded with a 5-point scale (Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). The Percentage of eyes with Grade 3 or higher was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0 | 0 | 0 | 0
  4-week Follow-up | 0 | 0 | 0 | 0

11. Primary Outcome: Corneal Neovascularization
Description: Corneal Neovascularization was assessed using a bio-microscope at baseline and 4- week evaluations in both eyes and was graded with a 5-point scale (Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). The Percentage of eyes with Grade 3 or higher was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0 | 0 | 0 | 0
  4-week Follow-up | 0 | 0 | 0 | 0

12. Primary Outcome: Corneal Staining
Description: Corneal Staining was assessed using a bio-microscope at baseline and 4- week evaluations in both eyes and was graded with a 5-point scale (Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). The Percentage of eyes with Grade 3 or higher was reported.
Time Frame: Baseline and 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0 | 0 | 0 | 0
  4-week Follow-up | 0 | 0 | 0 | 0

13. Primary Outcome: Tarsal Abnormalities
Description: Tarsal abnormalities were assessed using a biomicroscope at baseline, post lens fitting, 1-, 2- and 4- week evaluations in both eyes and was graded with a 5-point scale (Grade 0, 1, 2, 3 and 4) with grade 0 represents the absence of abnormalities and 1 to 4 representing successively worse abnormalities (i.e. Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). The percentage of eyes with Grade 3 or higher was reported.
Time Frame: 1-, 2- and 4-Week Follow-up
Population: The analysis population consists of all subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Subject Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  1-week Follow-up | 0 | 0 | 0 | 0
  2-week Follow-up | 0 | 0 | 0 | 0
  4-week Follow-up | 0 | 0 | 0 | 0

14. Primary Outcome: Percentage of Reported Ocular Symptoms (Cloudy/Blurry/Hazy)
Description: The Ocular symptom Cloudy/Blurry/Hazy was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 5.3 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 0.0

15. Primary Outcome: Percentage of Reported Ocular Symptoms (Dryness)
Description: The Ocular symptom Dryness was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 5.9 | 15.8 | 0.0 | 0.0
  4- Week Follow-up | 5.9 | 0.0 | 0.0 | 0.0

16. Primary Outcome: Percentage of Reported Ocular Symptoms (Grittiness/Foreign Body Sensation)
Description: The Ocular symptom Grittiness/Foreign Body Sensation was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 5.3 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 0.0

17. Primary Outcome: Percentage of Reported Ocular Symptoms (Irritation/Discomfort)
Description: The Ocular symptom Irritation/Discomfort was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 5.3 | 0.0 | 0.0
  4- Week Follow-up | 5.9 | 0.0 | 0.0 | 0.0

18. Primary Outcome: Percentage of Reported Ocular Symptoms (Itchiness/Scratchiness)
Description: The Ocular symptom Itchiness/Scratchiness was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 0.0 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 0.0

19. Primary Outcome: Percentage of Reported Ocular Symptoms (Lens Awareness)
Description: The Ocular symptom Lens awareness was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 10.5 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 0.0

20. Primary Outcome: Percentage of Reported Ocular Symptoms (Redness)
Description: The Ocular symptom Redness wasassessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 0.0 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 0.0

21. Primary Outcome: Percentage of Reported Ocular Symptoms (Variable Vision)
Description: The Ocular symptom Variable Vision was assessed by an individual item on a questionnaire and are subject reported, using the response scale of (N/A or Not recorded, Mild and rarely interferes with wear, Moderate and/or occasionally interferes with wear and Severe and/or frequently interferes with wear. The percentage of Moderate or severe symptoms were reported for the initial visit as well as the 1 month follow-up.
Time Frame: Baseline and 4-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Number analyzed (Participants) | 17 | 19 | 18 | 16
Number analyzed (Eyes) | 34 | 38 | 36 | 32
Percentage of Eyes
  Baseline | 0.0 | 0.0 | 0.0 | 0.0
  4- Week Follow-up | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 5 months.
Arm/Group | Etafilcon A | Prototype E1 | Prototype E2 | Prototype E3
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 1/19 | 4/19 | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etafilcon A (N=19) | Prototype E1 (N=19) | Prototype E2 (N=19) | Prototype E3 (N=19)
Non-significant Ocular Event (Eye disorders) | 1 (1) | 1 (1) | 4 (6) | 1 (1) — Includes Contact lens Papillary Conjunctivitis, Symptoms or Complaints requiring treatment, Slit lamp findings(Grade 2 or less) requiring treatment and using aosept solution to rinse lens resulting in burning and irritation.
Low Blood Pressure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not Study Related
Upset Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not Study Related
Muscle Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not Study Related
Minimal Skin Bruises (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not Study Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days